CLINICAL TRIAL: NCT00721318
Title: A Prevalence Study of Chronic Widespread Pain (CWP) Among Patients With Rheumatoid Arthritis (RA) and Control Population Matched by Gender, Age and Place of Residence in Tallinn and Harjumaa County
Brief Title: A Prevalence Study of Chronic Widespread Pain (CWP) Among Patients With Rheumatoid Arthritis (RA) and Control Population in Tallinn and Harjumaa County
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Estonian Society for Rheumatology (Other)
Responsible Party: Kati Otsa, MD, Estonian Society for Rheumatology
Other Study IDs: Merck35016; 35016
Record Dates: First submitted 2008-07-22; First posted 2008-07-24 (Estimated); Last update posted 2008-07-24 (Estimated); Status verified 2008-07

CONDITIONS: Chronic Widespread Pain
Keywords: chronic widespread pain; fibromyalgia; rheumatoid arthritis; Estonia
MeSH Terms: conditions — Chronic Pain; Fibromyalgia; Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Patients diagnosed with rheumatoid arthritis
- 2: Population controls to the subjects of group 1

SUMMARY:
The chronic widespread pain (CWP) and fibromyalgia (FM) cause serious discomfort, but at the same time they are not life threatening and they cannot be detected by any laboratory tests. The problems connected with these conditions have gained little attention in Estonia so far. It can be assumed that the CWP and FM often remain undetected and the sufferers live without treatment they need.

So far, there are no data on the prevalence of the CWP and FM in Estonia available.

The goal of the current research is to assess the prevalence of the CWP and local pain syndromes among Estonia's RA patients and among the control population in Tallinn and Harju County; also the factors connected with the presence of the pain and the pain treatment in use.

At the same time there will be a similarly designed research conducted in Jyväskylä Central Hospital, which provides the opportunity to compare results in Estonia's and Finland's research groups. The study on the distribution of the chronic pain among RA patients and control population will allow to assess the magnitude of the problem in Estonia and to raise the awareness of physicians about CWP and significance of its treatment.

Performing the study will provide an experience which forms the base for further epidemiological and clinical research on CWP and FM

ELIGIBILITY:
2000 RA patients from the East Tallinn Central Hospital's and the North Estonian Regional Hospital's in- and outpatients who live in Tallinn or Harju County

The control sample will be found from the Population Register through matching by gender, age (the same year) and place of residence (living in the city or in the countryside) with the subjects from RA sample according to the official procedure. If required, the research subjects from the control sample will be contacted by a rheumatologist participating in the study.

-

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Study population: Tallinn and Harju County (Estonia), population 552,000. The residents of both Tallinn and Harju County receive national health care services.
Sampling Method: Non-Probability Sample
Enrollment: 6000 (Estimated)
Dates: Start 2008-05; Primary Completion 2009-05 (Estimated); Study Completion 2010-05 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- East Tallinn Central Hospital, Tallinn, Estonia